CLINICAL TRIAL: NCT03903445
Title: Feasibility Study of the Masayang Pamilya Para sa Batang Pilipino (MaPa) Program From Families With Children and Adolescents
Brief Title: Masayang Pamilya Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ateneo de Manila University (Other)
Collaborators: University of Oxford (Other); University of Cape Town (Other); Philippines Department of Social Welfare and Development (Unknown); Philippines Child Protection Network (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AdMUREC_19_092PA
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Parent-Child Relations; Child Maltreatment; Child Behavior Problem; Parenting
Keywords: Parenting Program

STUDY DESIGN:
Intervention Model Description: Pre-post evaluation of 2 separate interventions (no comparison)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MaPa Kids (Experimental): Masayang Pamilya Para Sa Batang Pilipino Program (MaPa Kids) Parenting training for parents of children aged 2-9
  * Program length: 8 consecutive weekly sessions
  * Incentive: PHP 500 or approximately £7 per participant
  * Participants: N=15 per group
  Interventions: Behavioral: Masayang Pamilya Para Sa Batang Pilipino Program (MaPa Kids)
- MaPa Teens (Experimental): Masayang Pamilya Para Sa Tinedyer Pilipino Program (MaPa Teens) Parenting training for parents of children aged 10-17
  * Program length: 9 consecutive weekly sessions
  * Adult Incentive: PHP 500 or approximately £7 per participant
  * Child incentive: PHP 300 or approximately £4 per participant
  * Participants: N=15 per group
  Interventions: Behavioral: Masayang Pamilya Para Sa Tinedyer Pilipino Program (MaPa Teens)

INTERVENTIONS:
Behavioral: Masayang Pamilya Para Sa Batang Pilipino Program (MaPa Kids) — MaPa Kids is an 8-session parenting program delivered weekly to groups of parents (N=15 per group).
  The program includes the following content: 1) spending one-on-one time with children; 2) describing actions and feelings for cognitive development and socio-emotional awareness; 3) using praise and rewards to encourage positive behavior; 4) establishing limits through effective instruction giving and consistent household rules; 5) nonviolent discipline such as ignoring negative attention seeking behavior, and consequences for noncompliance, rule-breaking, and aggressive behavior; 6) problem solving with children; and 7) mindfulness based stress reduction.
  Other Names: Parenting for Lifelong Health for Young Children (PLH)
  Arms: MaPa Kids
Behavioral: Masayang Pamilya Para Sa Tinedyer Pilipino Program (MaPa Teens) — MaPa Teens is a 9-session parenting program delivered to groups of parents and children aged 10-17 (N=15 dyads per group).
  The program includes the following content: 1) one-on-one time with parents and teens, 2) positive reinforcement of positive behavior, 3) managing anger and stress, 4) establishing rules and routines, 5) family budgeting, 6) accepting responsibility for actions, 7) resolving family conflicts, 8) keeping safe in the community and resolving conflicts, and 9) reflection and moving on.
  Other Names: Parenting for Lifelong Health (PLH) for Adolescents
  Arms: MaPa Teens

SUMMARY:
The aim of this study is to test the feasibility of (1) an 8-session version of the Masayang Pamilya (MaPa) parenting program for families with children aged 2-9 (MaPa Kids) and (2) a culturally and contextually adapted 9-session MaPa parenting program for families with children aged 10-17 (MaPa Teens).

The feasibility of MaPa Kids and MaPa Teens will be assessed through self-report questionnaires, in-depth interviews and focus group discussions, and implementation data. Together, the focus groups, questionnaires, interviews, and implementation data will assess the overall feasibility of the MaPa Kids and MaPa Teen programs in the Philippines by examining program delivery, participation, acceptability, scalability, and preliminary effectiveness on reducing child maltreatment and associated risks.

DETAILED DESCRIPTION:
Child maltreatment occurs at much higher rates in low- and middle-income countries (LMIC) than in high-income countries. Parenting programs have shown particular promise in preventing child maltreatment, as well as improving child health and educational outcomes. However, there are currently very few parenting programs that are both evidence-based and affordable for LMIC, such as the Philippines, where the need is the greatest. For instance, the 2015 national baseline survey on violence against children (VAC) revealed that 80% of Filipino youth respondents had experienced violence in childhood, with 60% of these cases occurring at home. Mothers, fathers, and siblings were the most commonly reported perpetrators of harsh physical and psychological punishment (UNICEF, 2016). A logical recourse to decrease child maltreatment in the country is to implement interventions/programs that improve parents' relationships with their children and their knowledge and skills in child behavior management.

There is extensive scientific evidence that parenting support programs are effective in reducing child maltreatment and associated risk factors such as corporal punishment and parent negative psychological health (e.g., Desai, Reece & Shakespeare-Pellington, 2017; Mikton & Butchart, 2009). Parenting for Lifelong Health (PLH) is one such initiative led by UNICEF and WHO to support evidence-based parenting programs to reduce VAC in low and middle-income contexts.

In 2016-2017, PLH-Philippines embarked on the cultural adaptation, feasibility study (N=30), and pilot randomized control trial (RCT) (N=120) of the MaPa Kids program in the National Capital Region, which was implemented with families with children ages 2-6 and who were beneficiaries of the Department of Social Welfare and Development (DSWD) Pantawid Pamilyang Pilipino Program (4Ps). The results of this initial RCT were promising with reduced child maltreatment, dysfunctional parenting, less support of corporal punishment, lower levels of child problem behavior intensity, and higher sense of parenting efficacy at post-intervention reported by parents who participated in MaPa Kids compared to control group families who underwent the 4Ps Family Development Sessions (FDS). Reduced child maltreatment persisted at one-year follow-up assessment.

Building on the aforementioned trial, this study aims to expand the development, implementation, and evaluation of the parenting programs in the Philippines as part of a systematic effort to further assess the feasibility of (1) an 8-session version of the MaPa Kids program for families with children aged 2-9 and (2) a culturally adapted 9-session parenting program for families with children aged 10-17 (MaPa Teens).

The 8-session MaPa Kids and 9-session MaPa Teens modules will be piloted through a pre-post feasibility study. Both MaPa Kids and MaPa Teens parenting intervention modules will be implemented by eight local facilitators and two coaches in a low-income community - in Quezon City, Philippines - identified in collaboration with DSWD. Following participant recruitment and informed consent and assent procedures, baseline sociodemographic information and primary, proximal, and secondary information will be collected from parents/caregivers and their children (aged 10-17 in MaPa Teens).

Standardized baseline and one-month post-program questionnaires assessing primary and secondary outcomes, as well as demographic data, will be administered to 60 parents/primary caregivers and 30 children who participate in the program. Implementation data will be collected from parents/caregivers and program facilitators through report forms/checklists and video-recordings of each program session. Focus group discussions will be held with 60 parents/primary caregivers, 30 children aged 10-17, and eight program facilitators.

ELIGIBILITY:
Eligibility criteria Participants must have provided written, informed consent prior to the occurrence of any study procedures.

Inclusion criteria for participating parents or caregivers (N=60):

1. Age 18 or older;
2. Primary caregiver responsible for the care of a child between the ages 2-9 (Kids) or 10-17 (Teens);
3. Spend at least four nights a week in the same household as the child in the previous month;
4. Recipient of the 4Ps conditional cash transfer program;
5. Provision of consent to participate in the full study;
6. Provision of consent for their child to participate in the full study (for MaPa Teens only).

Exclusion criteria for adult parents:

1. Any adult who has already participated in the Parent Effectiveness Service;
2. Any adult exhibiting severe mental health problems or acute mental disabilities;
3. Any adult that has been referred to child protection services due to child abuse.

Inclusion criteria for child respondents (N=30):

1. Age 10 to 17 years at initial assessment;
2. Lives in the house at least 4 nights per week;
3. Must have an adult primary caregiver who lives in the household, who provides consent, and who participates in the study;
4. Provides assent to participate in the full study.

Exclusion criteria for child respondents:

1. Any child who is either experiencing severe mental health problems, has acute developmental disabilities and
2. If the child participant has been referred to social services during baseline data collection due to reported or observed indications of significant harm.

The study will also assess program fidelity and quality of delivery by program facilitators (N=8). These facilitators and coaches will have the following inclusion criteria:

1. Age 18 or older;
2. Prior participation in a 5-day facilitator training workshop;
3. Agreement to implement the entire program;
4. Provision of consent to participate in the full study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Child maltreatment of young children - physical and emotional abuse: ISPCAN Child Abuse Screening Tool-Trial Parent-Child Version (ICAST-TPC) - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Physical abuse and emotional abuse will be measured using items from an adapted and expanded version of the ISPCAN Child Abuse Screening Tool-Trial Parent version (ICAST-TP). The ICAST-T is an adaptation of the multi-national and consensus-based survey instrument ICAST-Parent version (ICAST-P), and has been used successfully in low and middle-income countries. The ICAST-TP measures parental reports of the incidence of abuse perpetrated against their child over the past month using a frequency score on a scale of 0 to 7, or 8 or more times (e.g., "In the past 4 weeks, how often did you discipline [Child Nickname] by pushing, grabbing, or kicking him/her?"). This study will assess incidence of child maltreatment for physical abuse (16 items), emotional abuse (10 items), as well as an overall indication of previous child abuse (0 = no abuse; 1 = previous abuse). We will also assess frequency of overall abuse by summing all of the subscales as well as for each individual subscale.
Child maltreatment of adolescents - physical and emotional abuse: ISPCAN Child Abuse Screening Tool-Trial Parent-Adolescent Version (ICAST-TPA) - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Physical and emotional abuse will be measured using items from an adapted and expanded version of the ISPCAN Child Abuse Screening Tool-Trial Parent version (ICAST-TP). The ICAST-T is an adaptation of the multi-national and consensus-based survey instrument ICAST-Parent version (ICAST-P), and has been used successfully in low and middle-income countries. The ICAST-TP measures parental reports of the incidence of abuse perpetrated against their child over the past month using a frequency score on a scale of 0 to 7, or 8 or more times (e.g., "In the past 4 weeks, how often did you discipline [Child Nickname] by pushing, grabbing, or kicking him/her?"). This study will assess incidence of child maltreatment for physical abuse (14 items), emotional abuse (10 items), as well as an overall indication of previous child abuse (0 = no abuse; 1 = previous abuse). We will also assess frequency of overall abuse by summing all of the subscales as well as for each individual subscale.
Child maltreatment of adolescents - physical and emotional abuse: ISPCAN Child Abuse Screening Tool-Trial Adolescent Version (ICAST-TA) - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Physical abuse (including abusive discipline) and emotional abuse will be measured using items from an adapted and expanded version of the ISPCAN Child Abuse Screening Tool-Trial Adolescent version (ICAST-TA). The ICAST-TA measures child reports of the incidence of abuse perpetrated against them over the past month using a frequency score on a scale of 0 to 7, or 8 or more times (e.g., "In the past 4 weeks, how often did your caregiver push, grab, or kick you?"). This study will assess incidence of child maltreatment for physical (10 items) and emotional (10 items), as well as an overall indication of previous child abuse (0 = no abuse; 1 = previous abuse). We will also assess frequency of overall abuse by summing all of the subscales as well as for each individual subscale.

SECONDARY OUTCOMES:
Child maltreatment of young children - physical abuse: ISPCAN Child Abuse Screening Tool-Trial Parent-Child Version (ICAST-TPC) - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Physical abuse (including abusive discipline) will be measured using 16 items from an adapted and expanded version of the ISPCAN Child Abuse Screening Tool-Trial Parent version (ICAST-TP). The ICAST-T is an adaptation of the multi-national and consensus-based survey instrument ICAST-Parent version (ICAST-P), and has been used successfully in low and middle-income countries, including recently in the Philippines. The ICAST-TP measures parental reports of the incidence of abuse perpetrated against their child over the past month using a frequency score on a scale of 0 to 7, or 8 or more times (e.g., "In the past 4 weeks, how often did you discipline [Child Nickname] by pushing, grabbing, or kicking him/her?").
Child maltreatment of young children - emotional abuse: ISPCAN Child Abuse Screening Tool-Trial Parent-Child Version (ICAST-TPC) - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Emotional abuse will be measured using 10 items from an adapted and expanded version of the ISPCAN Child Abuse Screening Tool-Trial Parent version (ICAST-TP). The ICAST-T is an adaptation of the multi-national and consensus-based survey instrument ICAST-Parent version (ICAST-P), and has been used successfully in low and middle-income countries, including recently in the Philippines. The ICAST-TP measures parental reports of the incidence of abuse perpetrated against their child over the past month using a frequency score on a scale of 0 to 7, or 8 or more times.
Child maltreatment of adolescents - physical abuse: ISPCAN Child Abuse Screening Tool-Trial Parent-Adolescent Version (ICAST-TPA) - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Physical abuse (including abusive discipline) will be measured using 14 items from an adapted and expanded version of the ISPCAN Child Abuse Screening Tool-Trial Parent version (ICAST-TP). The ICAST-T is an adaptation of the multi-national and consensus-based survey instrument ICAST-Parent version (ICAST-P), and has been used successfully in low and middle-income countries, including recently in the Philippines. The ICAST-TP measures parental reports of the incidence of abuse perpetrated against their child over the past month using a frequency score on a scale of 0 to 7, or 8 or more times (e.g., "In the past 4 weeks, how often did you discipline [Child Nickname] by pushing, grabbing, or kicking him/her?").
Child maltreatment of adolescents -emotional abuse: ISPCAN Child Abuse Screening Tool-Trial Parent-Adolescent Version (ICAST-TPA) - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Emotional abuse will be measured using 10 items from an adapted and expanded version of the ISPCAN Child Abuse Screening Tool-Trial Parent version (ICAST-TP). The ICAST-T is an adaptation of the multi-national and consensus-based survey instrument ICAST-Parent version (ICAST-P), and has been used successfully in low and middle-income countries, including recently in the Philippines. The ICAST-TP measures parental reports of the incidence of abuse perpetrated against their child over the past month using a frequency score on a scale of 0 to 7, or 8 or more times.
Child maltreatment - physical abuse: ISPCAN Child Abuse Screening Tool-Trial Adolescent Version (ICAST-TA) - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Physical abuse (including abusive discipline) will be measured using 10 items from an adapted and expanded version of the ISPCAN Child Abuse Screening Tool-Trial Adolescent version (ICAST-TA). The ICAST-TA measures child reports of the incidence of abuse perpetrated against them over the past month using a frequency score on a scale of 0 to 7, or 8 or more times (e.g., "In the past 4 weeks, how often did your caregiver push, grab, or kick you?"). This study will assess incidence of child maltreatment for physical (11 items).
Child maltreatment - emotional abuse: ISPCAN Child Abuse Screening Tool-Trial Adolescent Version (ICAST-TA) - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Emotional abuse will be measured using 10 items from an adapted and expanded version of the ISPCAN Child Abuse Screening Tool-Trial Adolescent version (ICAST-TA). The ICAST-TA measures child reports of the incidence of abuse perpetrated against them over the past month using a frequency score on a scale of 0 to 7, or 8 or more times.
Child neglect: ICAST-T Caregiver Neglect Subscale - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Child neglect will be assessed using an adapted version of the ICAST-T Caregiver (mentioned above) Neglect subscale. This subscale has three items for assessing medical, physical, and educational neglect, including "In the past month, how often was [Child Nickname] not taken care of when sick or injured, even when you or another caregiver were able to do so and could afford it?" and "In the past month, how often was [Child Nickname] not given a meal that he or she needed, even when you or another caregiver was able to afford it?"
Child neglect: ICAST-T Caregiver Neglect Subscale - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Child neglect will be assessed using an adapted version of the ICAST-T Caregiver (mentioned above) Neglect subscale. This subscale has five items for assessing medical, physical, and educational neglect, including "In the past month, how often was [Child Nickname] not taken care of when sick or injured, even when you or another caregiver were able to do so and could afford it?" and "In the past month, how often was [Child Nickname] not given a meal that he or she needed, even when you or another caregiver was able to afford it?"
Parental monitoring: Adapted Parental Monitoring Scale - Parent Report, MaPa Teens Only | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Parental monitoring and supervision practices will be measured using an adapted parental monitoring scale (11 items) which scale measures parents' solicitation of information (5 items, i.e., "How much do you try to know…") concerning their child's activities and friendships (e.g., who your child spends time with) using a 3-point scale (0 = I don't try; 2 = I try a lot); rule-setting, or how often parents set rules or limits about the same items using a 4-point scale (0 = Never; 3 = Always). Three items on monitoring online activities were added to the solicitation of information subscale (e.g., "How much do you try to know the websites your child visits?) and two items were added to the rule-setting subscale (e.g., "How much do you set rules or limits on how long your child uses his or her device?), derived from the Global Kids Online survey. Mean scores on the subscales are standardized and summed to create a parental monitoring score.
Parental monitoring: Adapted Parental Monitoring Scale - Child Report, MaPa Teens Only | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Parental monitoring and supervision practices will be measured using an adapted parental monitoring scale (20 items). The scale measures parents' solicitation of information (7 items, i.e., "How much do you try to know…") concerning their child's activities and friendships (e.g., who your child spends time with) using a 3-point scale (0 = I don't try; 2 = I try a lot); rule-setting, or how often parents set rules or limits about the same items using a 4-point scale (0 = Never; 3 = Always). Four items on monitoring of online activities were added to the solicitation of information subscale (e.g., "How much do you try to know the websites your child visits?) and nine items were added to the rule-setting subscale (e.g., "How much do you set rules or limits on how long your child uses his or her device?), derived from the Global Kids Online survey. Mean scores on the two subscales are standardized and summed to create a total parental monitoring score.
Child behavior problems: Child and Adolescent Behavior Inventory (CABI) - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Child behavior problems will be measured using the Child and Adolescent Behavior Inventory (CABI) (14 items). The CABI assesses a wide range of internalizing and externalizing symptoms in children and adolescents and is relatively shorter than the Child Behavior Check List (CBCL), making it a practical and reliable tool for measuring behavior problems. Parents report on their child's behavior during the past month (0 = Not True, 1 = Somewhat or Sometimes True, 1 = Very True). The irritability subscale (4 items, e.g., "has frequent mood changes") and the externalizing subscale (10 items, e.g., often lies or cheats) will be used to measure problem behaviors. Items on both subscales are summed to create a total score of child behavior problems.
Child behavior problems: Child and Adolescent Behavior Inventory (CABI) - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Child behavior problems will be measured using the Child and Adolescent Behavior Inventory (CABI). The CABI assesses a wide range of internalizing and externalizing symptoms in children and adolescents and is relatively shorter than the Child Behavior Check List (CBCL), making it a practical and reliable tool for measuring behavior problems. Children report on their own behavior during the past month (0 = Not True, 1 = Somewhat or Sometimes True, 1 = Very True). The irritability subscale (4 items, e.g., "has frequent mood changes") and the externalizing subscale (10 items, e.g., often lies or cheats) will be used to measure problem behaviors. Items on both subscales are summed to create a total score of child behavior problems.
Three Problem Rating Scale - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  The Three Problem Scale-Child Report (6 items) specific concerns or issues parents are having with their children change during an intervention. Parent-defined concerns from the Three Problem Scale that is consistent or larger than other measurements such as the Strengths and Difficulties Questionnaire or Child Behavior Check List. This study adapted the parent-report scale for children to report on specific issues or problems they are having with their parents. Children are asked to identify up to 3 areas of conflict with their parents that are causing them the most distress and to rate each problem area from 1 to 10 (1 = "not a problem," 10 = "couldn't be worse"). The same problem areas are then asked at post-assessment to assess whether these problems have changed. Each single item will be analysed separately as well as a total problem rating score for the 3 issues.
Three Problem Rating Scale - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  The Three Problem Scale-Parent Report (9 items) was adapted from developed by Scott to assess whether specific concerns or issues parents are having with their children change during an intervention. Parent-defined concerns from the Three Problem Scale that is consistent or larger than other measurements such as the Strengths and Difficulties Questionnaire or Child Behavior Check List. Parents are asked to identify up to 3 areas of concern with their children that are causing them the most distress and to rate each problem area from 1 to 10 (1 = "not a problem," 10 = "couldn't be worse"). The same problem areas are then asked at post-assessment to assess whether these problems have changed. Each single item will be analysed separately as well as a total problem rating score for the 3 issues.
Parenting efficacy: Parenting Sense of Competence Scale (PSOC-ES) - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Parenting efficacy will be assessed using the Efficacy Subscale of the Parenting Sense of Competence Scale (8 items; PSOC-ES). The PSOC has been widely used in studies to evaluate parenting self-esteem, efficacy, or competence. The PSOC Efficacy Subscale measures parental perception of competence, problem-solving ability, and capability in the parenting role (e.g., "I honestly believe I have all the skills necessary to be a good mother/father to my child"). Each item is rated on a 6-point scale that ranges from 1 (strongly disagree) to 6 (strongly agree). Items are summed to create a total score of parental self-efficacy.
Parenting stress: Parental Stress Scale (PSS) - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Parenting stress will be assessed using the Parental Stress Scale (PSS; 18 items). PSS has been widely used to measure parenting stress, including in LMIC, such as Pakistan and China. The scale has also been used with non-parent caregivers such as grandparents. Caregivers report current positive attitudes (n = 8, e.g., "I feel close to my child") and negative attitudes (n = 10, e.g., "I feel overwhelmed by the responsibility of being a parent") related to parenting stress based on a five-point Likert scale (0 = strongly disagree; 4 = strongly agree). Positive items are reversed and then all items are summed to create a total parenting stress score (range 0 to 90).
Self-efficacy in managing emotions - Regulatory Emotional Self-Efficacy Scale - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Self-efficacy in managing emotions is measured using an adapted version of the Regulatory Emotional Self-Efficacy Scale (8 items). The anger-irritation subscale includes four items. Parents indicate how well they think they can control their emotions (e.g., How well can you manage negative feelings when reprimanded by significant others?) using a 5-point scale (1 = Not well at all to 5 = Very well). Scores are averaged to create a total score for self-efficacy in managing emotions.
Parental depressive symptoms - Moods and Feelings Questionnaire (MFQ) - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Parental depressive symptoms will be measured using the adult version of Moods and Feelings Questionnaire (MFQ). The scale includes 13 items indicating depressive symptoms (e.g., I didn't enjoy anything at all). Parents indicate how they have been feeling or acting in the past two weeks using a 3-point Likert scale (0 = Not true, 1 = Sometimes True, 2 = True). Items are summed to create a total parental depression score.
Child depressive symptoms - Moods and Feelings Questionnaire (MFQ) - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Child depressive symptoms will be measured using the short parent report version of Moods and Feelings Questionnaire (MFQ). The scale includes 13 items indicating depressive symptoms (e.g., I didn't enjoy anything at all). Parents indicate how their child has been feeling or acting in the past two weeks using a 3-point Likert scale (0 = Not true, 1 = Sometimes True, 2 = True). Items are summed to create a total child depressive symptoms score.
Child depressive symptoms - Moods and Feelings Questionnaire (MFQ) - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Child depressive symptoms will be measured using the short child report version of Moods and Feelings Questionnaire (MFQ). The scale includes 13 items indicating depressive symptoms (e.g., I didn't enjoy anything at all). Children indicate how they have been feeling or acting in the past two weeks using a 3-point Likert scale (0 = Not true, 1 = Sometimes True, 2 = True). Items are summed to create a total child depressive symptoms score.
Parent exposure to intimate partner violence and intimate partner coercion - Revised Conflict Tactics Scale Form (CTS2S) - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Adult self-report of experiencing intimate partner violence over the past month will be assessed using an adapted version of the Revised Conflict Tactics Scale Short Form (CTS2S, 8 items). The CTS2S includes 2 items on the frequency of negotiation (e.g., "partner suggested a compromise for a disagreement"), 5 items on physical assault (e.g., "partner pushed, shoved, or slapped me"), and 1 item on psychological aggression (e.g., "partner insulted, shouted, yelled, or swore at me").
Parent exposure to intimate partner violence and intimate partner coercion - WHO Multi-Country Study Questionnaire- Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Adult self-report of experiencing intimate partner violence over the past month will be assessed using adapted items from the WHO Multi-Country Study Questionnaire on Women's Health and Life and Domestic Violence against Women (WHO, 10 items). The adapted WHO questionnaire includes 7 items on coercion and emotional violence (e.g., "my partner tried to keep me from seeing my friends" and "my partner insisted on knowing where I was at all times"), and 3 items on restriction of financial autonomy (e.g., "my partner took my earnings or savings from me against my will.") All answers are coded on a frequency scale of 0 to 3 (0 = never happened; 1 = once or twice; 2 = 3-5 times; 3 = more than 5 times). Both the CTS2S and the WHO will determine an overall indication of intimate partner violence on a level of severity (sum of items across both scales) and prevalence (dichotomous variable indicating experience of conflict or not), as well as for each subscale.
Family functioning - Burmese Family Functioning Scale - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Family functioning will be measured using the Burmese Family Functioning Scale. It includes subscales on family cohesion (12 items, e.g., having understanding towards one another), family communication (7 items, e.g., expressing love through words or actions), and negative family interactions (4 items, e.g., having a lot of bad feelings in the family). Parents indicate how much they agree with statements regarding their family in the last four weeks on a 4-points Likert scale (1 = Almost Never True; 4 = Almost Always True). Items are summed to create total frequency score as well as for each subscale.
Family functioning - Burmese Family Functioning Scale - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Family functioning will be measured using the Burmese Family Functioning Scale. It includes subscales on family cohesion (12 items, e.g., having understanding towards one another), family communication (7 items, e.g., expressing love through words or actions), and negative family interactions (4 items, e.g., having a lot of bad feelings in the family). Children indicate how much they agree with statements regarding their family in the last four weeks on a 4-points Likert scale (1 = Almost Never True; 4 = Almost Always True). Items are summed to create total frequency score as well as for each subscale.
Community violence exposure: Violence Exposure Scale - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Exposure to community violence will be measured using 6 items from each of the subscales of the Violence Exposure Scale: Witnessing Community Violence and Experiencing Community Violence (12 items total). Parents report on whether they witnessed or experienced community violence in the past month based on 4-point Likert scale (0 = never; 4 = Often, more than 5 times). They also have the option to report that the incident has occurred before but not in the past month. Items from each subscale are summed to create a total subscale score as well as to create an incidence rating of exposure to community violence.
Community violence exposure: Violence Exposure Scale - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Exposure to community violence will be measured using 6 items from each of the subscales of the Violence Exposure Scale: Witnessing Community Violence and Experiencing Community Violence (12 items total. Children report on whether they witnessed or experienced community violence in the past month based on 4-point Likert scale (0 = never; 4 = Often, more than 5 times). They also have the option to report that the incident has occurred before but not in the past month. Items from each subscale are summed to create a total subscale score as well as to create an incidence rating of exposure to community violence.
Positive parenting: Parenting of Young Children Scale (PARYC) - Parent Report, MaPa Kids Only | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Positive parenting behavior will be assessed using the Parenting of Young Children Scale (PARYC, 21 items). The PARYC measures the frequency of parent behavior over the previous month. Items are summed to create total frequency scores for positive parenting (7 items, e.g., "how often do you play with your child"), setting limits (7 items, e.g., "how often do you stick to your rules and not change your mind") and proactive parenting (7 items, e.g., "how often do you explain what you want your child to do in clear and simple ways"). It has been used with strong reliability in previous studies on the program adapted in this study.
Dysfunctional parenting: Parenting Scale (PS) - Parent Report, MaPa Kids Only | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Dysfunctional parenting behavior will be assessed using the Parenting Scale (PS, 30 items). This scale examines parent attitudes and beliefs regarding discipline practice. Responses are based on a 7-point Likert scale in which parents are presented with a situation and then are asked to choose between two alternative responses to a situation (1 = most effective; 7 = most ineffective; i.e., situation: "When I say my child can't do something;" response, score = 1: "I stick to what I said;" or response score = 7: "I let my child do it anyway"). Items are summed to create an overall score as well as for three subscales: Laxness, Over-reactivity, and Verbosity. The PS has been used widely to assess the effectiveness of parenting programs, including in low-resource settings such as Panama.
Parenting behavior: Alabama Parenting Questionnaire - Parent Report, MaPa Teens Only | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Parent-child interaction, will be measured using two subscales from the Alabama Parenting Questionnaire - Adult Report: Positive Parenting (8 items, e.g., "you praise your child if s/he behaves well") and Parent Involvement (8 items, e.g., "you take your child to a special activity"). The APQ has been shown to have moderate to strong internal reliability for both parent and child reports (Cronbach's alpha = 0.50 to 0.89). It has been used widely including in LMIC such as South Africa and Mexico. Caregivers report on the frequency of parenting behavior based on a 4-point Likert scale (0 = never; 3 = Often, more than 5 times). Items are summed to create total frequency score (range 0 to 24) as well as for each subscale.
Parenting behavior: Alabama Parenting Questionnaire - Child Report, MaPa Teens Only | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Parent-child interaction, will be measured using two subscales from the Alabama Parenting Questionnaire - Child Report: Positive Parenting (8 items, e.g., "your parent/caregiver praises you when you behave well") and Parent Involvement (9 items, e.g., "your parent/caregiver takes you child to a special activity"). The APQ has been shown to have moderate to strong internal reliability for both parent and child reports (Cronbach's alpha = 0.50 to 0.89). It has been used widely including in LMIC such as South Africa and Mexico [31-36]. Caregivers report on the frequency of parenting behavior based on a 4-point Likert scale (0 = never; 3 = Often, more than 5 times). Items are summed to create total frequency score (range 0 to 24) as well as for each subscale.
Attitudes toward punishment: UNICEF Multiple Indicator Cluster Survey (MICS) 5 Child Discipline Module - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Attitudes toward punishment will be assessed using one item from the UNICEF Multiple Indicator Cluster Survey (MICS) 5 Child Discipline module. The MICS item asks the parent/primary caregiver: "In order to bring up, raise up, or educate a child properly, the child needs to be physically punished." Parents/primary caregivers will report whether they disagree or agree with the statement based on a 5-point Likert scale of 0 to 4 (0 = Disagree strongly; 4 = Agree strongly).
Attitudes toward punishment: UNICEF Multiple Indicator Cluster Survey (MICS) 5 Child Discipline Module - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Attitudes toward punishment will be assessed using one item from the UNICEF Multiple Indicator Cluster Survey (MICS) 5 Child Discipline module
Attitudes towards punishment: ISPCAN Child Abuse Screening Tool-Intervention and Efficacy and Attitudes Sub-Scales - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Attitudes toward punishment will be assessed using items from each of the ISPCAN Child Abuse Screening Tool-Intervention Efficacy and Attitudes sub-scales (ICAST-I). The two ICAST-I Efficacy items asks how often parents/primary caregivers reacted to child misbehavior over the past month using a frequency score on a scale of 1 to 7, or 8 or more times (e.g., "In the past 4 weeks, how often did physical discipline seem like the only option for stopping [Child Nickname's] bad behavior?". Four of the ICAST-T Attitudes sub-scale items assess parent/primary caregiver refer to a scenario in which a child is "always getting into trouble," and asks about the level of effectiveness of various disciplinary responses based on a 5-point Likert scale of 1 to 5 (1 = Very ineffective; 5 = Very effective). The fifth item on this sub-scale then asks "Which of the above approaches do you feel is most effective for disciplining children?" and permits a single select response.
Attitudes towards punishment: ISPCAN Child Abuse Screening Tool-Intervention and Efficacy and Attitudes Sub-Scales - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Attitudes toward punishment will be assessed items from the ISPCAN Child Abuse Screening Tool-Intervention Efficacy and Attitudes sub-scales (ICAST-I). Four of the ICAST-T Attitudes sub-scale items refers to a scenario in which a child is "always getting into trouble," and asks about the level of effectiveness of various disciplinary responses based on a 5-point Likert scale of 1 to 5 (1 = Very ineffective; 5 = Very effective). The fifth item on this sub-scale then asks "Which of the above approaches do you feel is most effective for disciplining children?" and permits a single select response.
Child prosocial behavior: Prosocial Behavior Scale - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Child prosocial behavior will be measured using a Prosocial Behavior Scale. Children report how often they engage in prosocial behaviors (16 items, e.g., "I share things I have with my friends") using a 5-point Likert Scale (0 = Never/Almost Never; 5 = Almost Always/Always True). Items are averaged to create a total score for child prosocial behavior.
Child risk behavior: Risk Behavior Scale - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Child risk behavior will be measured using a Risk Behavior Scale. Children report how many times they have engaged in risky behaviors in the past month (8 items, e.g., "drinking beer or wine") using a using a frequency score on a scale of 0 to 7, or 8 or more times. Items are summed to create a total score for child risk behavior. This measure will be administered using audio-CASI to increase response rate.
Witnessing family violence: ICAST-T Child - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  The incidence and frequency of witnessing family violence will be assessed by using two items from the ICAST-T Child (e.g., "How many days in the past month were there arguments with adults shouting in your home?"). Items will be summed to create a total frequency of witnessing family violence as well as dichotomized to create an incidence variable.
Parental Support for School - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Parental support for school will be measured by asking how often the parent engages in behaviours that support learning (6 items) using a 5-point Likert scale. Higher scores reflect more parental support and value for school.
Parental Support for School - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Parental support for school will be measured by asking how often the parent engages the child in behaviours that support learning (6 items) using a 5-point Likert scale. Higher scores reflect more parental support and value for school.
Educational Aspirations - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Educational aspirations will be measured one item asking the parent "How far would like your child to go in school?" rated on a 5-point scale (1 = finish some high school, 2 = graduate from high school, 3 = graduate from a 2-year college, 4 = graduate from a 4-year college, 5 = graduate from law, medical or graduate school).
Educational Aspirations - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Educational Aspirations will be measured one item asking the child "How far would you to go in school?" rated on a 5-point scale (1 = finish some high school, 2 = graduate from high school, 3 = graduate from a 2-year college, 4 = graduate from a 4-year college, 5 = graduate from law, medical or graduate school).
Educational Expectations - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Educational Expectations will be measured using one item asking the parent how far they think their child will actually go in school rated on the same 5-point scale (1 = finish some high school, 2 = graduate from high school, 3 = graduate from a 2-year college, 4 = graduate from a 4-year college, 5 = graduate from law, medical or graduate school).
Educational Expectations - Child Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Educational Expectations will be measured using one item asking the child how far they think they will actually go in school rated on the same 5-point scale (1 = finish some high school, 2 = graduate from high school, 3 = graduate from a 2-year college, 4 = graduate from a 4-year college, 5 = graduate from law, medical or graduate school).

OTHER OUTCOMES:
Recruitment rate | Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Number of families who were eligible for inclusion and provided consent to participate in the program divided by the number of target population who were exposed to recruitment activities
Enrollment rate | Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Number of families who attend at least one session of the program divided by the number of families recruited into the program
Participation rate | Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Mean attendance rate for program sessions based on those families who enrolled in the program (i.e., parents who attended at least one session). Percentage of families who enrolled in the program who attended 50% (e.g., 6 sessions) and 75% (e.g., 9 sessions) or more.
Implementation Dosage in hours | Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Average number of hours delivered by facilitators (time for pre-program consultation plus session plus phone consultations per participant, facilitator report verified by implementation monitors).
Implementation Dosage (points of contact) | Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Total number of points of contact by facilitators.
Implementation Fidelity (percentage of session activities delivered per session) | Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Percentage of number of session activities delivered by facilitators (by facilitator group, implementing agency, and participating country site; facilitator fidelity check-list reports verified by implementation monitors and random video recordings of session delivery)
Implementation Fidelity (mean percent of activities delivered per session) | Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Average number of activities delivered divided by total number of activities per session (by facilitator group, implementing agency, and participating country site; facilitator reports verified by implementation monitors and random video recordings of session delivery)
Implementation Quality | Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  The implementation quality is assessed using the PLH-Facilitator Assessment Tool (PLH-FAT): Seven standard behaviour categories are grouped into two scales based on the core activities and process skills. Assessment of core activities includes quality of delivery during home activity review, illustrated story discussions, and practicing skills with scores from 0 (inadequate) to 3 (exceeds expectations). Assessment of process skills includes modelling skills, collaborative facilitation approach, encouragement of participation, and leadership skills (scoring from 0 = inadequate to 3 = outstanding). The total scores oft both subscales range from 0 to 72 with higher scores indicating higher facilitator competency. The total percent score for both subscales will be calculated (total score / total possible score) x 100%. A higher percent score indicates higher implementation quality.
Participants observed change in parenting practices and child behaviour at home during program | Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Focus groups with participants and facilitators in order to explore program acceptability.
Existing barriers to participation during sessions and engagement in home practice and other activities | Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Focus groups with participants and facilitators in order to explore program acceptability.
Challenges in implementing the program | Post (approx. 1 month after end of intervention, i.e., 4 months post pre-assessment)
  Qualitative focus group discussions with the facilitators exploring challenges in implementing the program on a process (e.g., using a collaborative approach and/or explaining concepts such as child led play) and logistical level (e.g., recruitment, session length, location, meals).
Basic caregiver and child demographic information | Baseline
  Basic caregiver and child demographic information will be asked using items from the UNICEF Multiple Indicators Cluster Survey (MICS) Household Survey. The MICS was developed to monitor the situation of children and women on a global level and is based on Demographic and Health Surveys. It has been used widely throughout low- and middle-income countries (LMIC) including the Philippines. It assesses caregiver/child age, gender, marital status, employment status, education level, basic literacy, child's relationship to caregiver, presence of child's biological parents (including reasons for absence), and other household members' age, gender and relationship to caregiver. It also assesses other household socio-demographic characteristics including household structure, family employment, and whether or not the family receives any government grants
Household ladder - Parent Report | Baseline
  Subjective social status will be assessed using the MacArthur Subjective Scale of Social Status. Parents will be presented with a drawing of a 10-rung ladder that represents where people stand in their communities. The top of the ladder represents the highest standing in the community and the bottom ladder represents the lowest standing in their community. They will be asked to place themselves on the rung that best represents where they see themselves relative to their community (1 = lowest standing to 10 = highest standing).
Household income - Parent Report | Baseline
  An objective measure of household income will be obtained by asking parents to indicate their family's monthly income using a 16-item scale with income ranges from 0 = no income to 15 = over 83,000 monthly.
Adult history of child maltreatment - Parent Report | Baseline
  Parental/primary caregiver history of experiencing child maltreatment will be measured using an adapted ISPCAN Child Abuse Screening Tools Retrospective version (ICAST-R) (3 items). This scale utilizes parental self-reports of experiences during childhood (until age 18) to assess the history of ever experiencing physical (e.g., "When you were growing up (before age 18), did your caregiver ever discipline or punish you physically by hitting, spanking, slapping, kicking, or shaking you?") and emotional abuse (e.g., When you were growing up (before age 18) did any person ever discipline or punish you by insulting or criticizing you, to make you feel that you were bad, stupid or worthless?") (2 items). In this study, ever experiencing physical or emotional abuse will be assessed on a frequency scale (0 = Never; 1 = Once or twice; 2 = 3-5 times; 3 = More than 5 times). There will also be a dichotomous score for overall indication of previous child abuse (0 = no abuse; 1 = previous abuse).
Basic necessities - Parent and Child Report | Baseline
  Relative poverty will be assessed using the Basic Necessities Scale (8 items). Developed by the Center for South African Social Policy in the 'Indicators of Poverty and Social Exclusion Project,' the Basic Necessities Scale measures levels of economic deprivation by identifying basic household items that families are unable to afford. These include food, toiletries, clothes, shoes, and school uniforms, equipment, and fees. Items are coded dichotomously for positive or negative responses and summed to create an overall score. Previous studies in have used this scale in multiple settings with high internal reliability (alpha = .84). This information will be collected from both children and caregivers.
Household hunger - Parent Report | Baseline
  Relative poverty will be based on household hunger assessed using the Hunger Scale Questionnaire. This scale examines food shortage and hunger in the household. Parents respond positively or negatively regarding the occurrence of hunger in the household, whether it occurred during the past 30 days, and if so, whether it occurred more than 5 times in the past 30 days (e.g., "the household has run out of money to buy food"). The scale produces scores for single occurrence and intensity of hunger.
Food consumption - Parent Report | Baseline
  This study will also assess food consumption via caregiver report on average meals consumed per day in the past week for both the caregiver and child participants based on items from the UNICEF MICS Household Survey (e.g., "how many meals did you consumer per day").
Caregiver alcohol use - Parent Report | Baseline
  Parental dependency on alcohol will be assessed by assessing alcohol consumption during the past month (1 item). Dependency is based on 3 or more drinks per day for female participants and 5 or more per day for male participants. Due to the sensitive nature of these items, additional items dealing with other activities to reduce stress have been included in this section to encourage accuracy (3 items; e.g., "In the past month, have you been for a walk or done some other exercise to help you relax?").

CONTACTS AND LOCATIONS:
Overall Officials: Rosanne Jocson, PhD, Principal Investigator — Ateneo de Manila University; Liane P Alampay, PhD, Principal Investigator — Ateneo de Manila University; Jamie M Lachman, DPhil, Principal Investigator — University of Oxford; Frances Gardner, DPhil, Principal Investigator — University of Oxford; Engels Del Rosario, Principal Investigator — Department of Social Welfare and Development, Philippines; Bernadette Madrid, PhD, Principal Investigator — Child Protection Network, Philippines; Catherine L Ward, PhD, Principal Investigator — University of Cape Town
Locations (1):
- Ateneo de Manila University, Quezon City, Philippines

IPD SHARING:
Plan to Share IPD: Yes
It is planned to share results of this study to members of the scientific community with an interest in parenting interventions and process evaluation. The aim is to sustain the intervention after the end of the project. Following the analyses, all participant data will be de-identified and stored using the United Kingdom Archive Standards (www.data-archive.ac.uk/create-manage/planning-for-sharing). Anonymized data will also be included as secondary data in SUPER (Scale-Up of Parenting Evaluation Research).
  Supporting Information: Study Protocol
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the primary papers from the study have been published, all participant data will be de-identified and stored indefinitely using United Kingdom Data Archive standards (www.data-archive.ac.uk/create-manage/planning-for-sharing).
Access Criteria: Following the data analyses from the feasibility pilot, all participant data will be de-identified and stored using United Kingdom Data Archive standards (www.data-archive.ac.uk/create-manage/planning-for-sharing). De-identification will include removal of direct identifiers (names, addresses, postcode information, telephone numbers or pictures) as well as indirect identifiers (information on location, occupation or any other information that could be linked to a public source). This will include removing or aggregating variables or reducing the precision or detailed textual meaning of a variable in the dataset. Access to this data will be controlled and require authorisation from the research team for further use.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-31): https://cdn.clinicaltrials.gov/large-docs/45/NCT03903445/Prot_SAP_000.pdf